CLINICAL TRIAL: NCT02137395
Title: The Effect of Dexamethasone on Sugammadex Reversal in Pediatric Patients Undergoing Adenotonsillectomy: a Randomized, Placebo-controlled Study
Brief Title: The Effect of Dexamethasone on Sugammadex Reversal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ersel GULEC, Assist.Prof., Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DXSX01
Record Dates: First submitted 2014-05-12; First posted 2014-05-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Incomplete Reversal of Neuromuscular Block
Keywords: Children, Dexamethasone, Sugammadex,
MeSH Terms: interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Experimental): Patients are received dexamethasone via intravenous (iv) route of 0.5 mg.kg-1 (maximum dose of 8 mg) in group D at the induction of anesthesia.
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): An equal volume of saline iv in group S at the induction of anesthesia.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — dexamethasone administration, intravenously
  Other Names: Dekort
  Arms: Dexamethasone
Drug: Placebo — saline administration intravenously
  Other Names: Saline,0.9% NaCl
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether dexamethasone extends the duration of recovery from anesthesia.

DETAILED DESCRIPTION:
After obtaining Local Ethics Committee of Cukurova University approval and written parental consent, this prospective, randomized, double blind, placebo-controlled study will be performed. Sixty patients scheduled for elective tonsillectomy or adenoidectomy, aged 3-8 years with American Society of Anesthesiologists physical status 1 and 2 are recruited to the study. Exclusion criteria are the presence of respiratory, hepatic, renal and cardiovascular disease, oropharyngeal or facial pathology, neuromuscular disorder, hypertension and diabetes mellitus. Patients are randomly allocated into two groups in a 1:1 ratio by a computer-generated list. Allocation is provided with sealed envelopes containing group named paper.

Patients are admitted to the preoperative unit 30 minutes before the operation. All patients are monitored with non-invasive blood pressure (NIBP), electrocardiogram (ECG), end-tidal carbon dioxide (ETCO2) and peripheral oxygen saturation (SpO2) in the operating room before the start of anesthesia induction. Anesthesia is induced with 4-5 % sevoflurane and a cannula (18 gauges) is placed intravenously after ensuring adequate depth of anesthesia and thus 0.9% of saline infusion is started at a 10 mL kg-1 hr-1 rate for hydration. Patients are received dexamethasone via intravenous (iv) route of 0.5 mg.kg-1 (maximum dose of 15 mg) and an equal volume of saline iv, in group D and group S, respectively.

Neuromuscular monitoring is initiated after the induction of anesthesia by an acceleromyograph (TOF-Watch® S; Organon Ireland Ltd, Drynam Road, Swords, Co. Dublin, Ireland) measuring the function of adductor pollicis muscle. A transducer is attached over the thumb. Two electrodes are placed on cleaned skin corresponding to the ulnar nerve trajectory at the wrist. Stabilization and calibration are performed for TOF-Watch S according to good clinical research practice in pharmacodynamic studies of NMBAs. (Fuchs-Buder, Claudius et al. 2007) After calibration, Train of Four stimulations (TOF) are applied repetitively every 15 minutes for 3 minutes. Rocuronium is administered intravenously at a dose of 0.6 mg.kg-1 followed by calibration period. Tracheal intubation is performed after obtaining the adequate neuromuscular blockade. TOF stimulation is maintained every 15 minutes until the end of anesthesia, or until the TOF ratio is 0.9. SpO2, ECG and NIBP monitoring with 10 minutes intervals and neuromuscular data obtained by TOF-Watch® S are recorded. When the T2 of the TOF reappeared, all patients are administered a single bolus injection of sugammadex at a dose of 2 mg.kg-1. The time to achieve a TOF ratio of 0.9 after sugammadex administration is recorded for all patients.

At the end of surgery anesthesia is terminated and the awake patients are extubated. After extubation, patients are transported to the postoperative care unit. Pulse oximetry, respiratory rate and non-invasive blood pressure monitoring, the level of consciousness and clinical evaluation of recovery (5 s head lift test, absence of diplopia, tongue depressor test, and general muscle weakness) are recorded with 15 minutes intervals during 60 minutes in the postanesthesia care unit (PACU). Any adverse effects are recorded during the surgery and postoperatively for 10 hours. All records and drug administrations are performed by an anesthetist, who is blinded to the patient group. The primary endpoint is defined as the time to achieve TOF ratio to 0.9 after sugammadex administration.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective tonsillectomy or adenoidectomy,
* aged 3-8 years
* with American Society of Anesthesiologists physical status 1 and 2

Exclusion Criteria:

* the presence of respiratory, hepatic, renal and cardiovascular disease,
* oropharyngeal or facial pathology
* neuromuscular disorder
* hypertension
* diabetes mellitus.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the time to achieve TOF (Train of Four stimulation) ratio to 0.9 after sugammadex administration. | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ersel Gulec, M.D., Principal Investigator — Cukurova University Faculty of Medicine
Locations (1):
- Cukurova University Faculty of Medicine, Adana, Turkey (Türkiye)

REFERENCES:
- [Result] Rezonja K, Sostaric M, Vidmar G, Mars T. Dexamethasone produces dose-dependent inhibition of sugammadex reversal in in vitro innervated primary human muscle cells. Anesth Analg. 2014 Apr;118(4):755-63. doi: 10.1213/ANE.0000000000000108. PMID 24651229
- [Result] Plaud B, Meretoja O, Hofmockel R, Raft J, Stoddart PA, van Kuijk JH, Hermens Y, Mirakhur RK. Reversal of rocuronium-induced neuromuscular blockade with sugammadex in pediatric and adult surgical patients. Anesthesiology. 2009 Feb;110(2):284-94. doi: 10.1097/ALN.0b013e318194caaa. PMID 19194156